CLINICAL TRIAL: NCT00581113
Title: A Study of Neural Stem Cell (NSC) Preserving Whole Brain Radiation Therapy (WBRT) and Stereotactic Radiosurgery in Patients With 1-6 Brain Metastases
Brief Title: Neural Stem Cell Preserving Brain Radiation Therapy & Stereotactic Radiosurgery in Patients With 1-6 Brain Metastases
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: New research priorities
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-10655
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Lung Cancer; Breast Cancer; Prostate Cancer
Keywords: whole brain radiotherapy; neural stem cell; brain metastases; radiosurgery
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Brain Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard Whole Brain Radiotherapy
  Interventions: Radiation: Radiotherapy
- 2 (Experimental): Neural Stem Cell-Preserving Whole Brain Radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Treatments are delivered through parallel opposed or 5 degree RAO/LAO fields that cover the entire cranial contents. There should be beam fall-f of at least 1 cm. The eyes must be excluded from the beam either by field arrangement or shielding.

SUMMARY:
For patients with 1-6 intraparenchymal brain metastases from various primary histologies (except for melanoma), stereotactic radiosurgery (administered upfront or concurrently) or complete surgical resection with neural stem cell (NSC)-preserving whole-brain radiotherapy (WBRT) results in improved neurocognitive profile over standard WBRT. The goal of this study is to assess feasibility of this treatment approach.

DETAILED DESCRIPTION:
Cancer patients (except patients with melanoma) with 1-6 brain metastases are randomized to receive standard whole brain radiation therapy or whole brain radiation therapy in a neural stem cell-preserving manner.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-melanoma primary malignancy with 1-6 intraparenchymal brain metastases (or small cell lung cancer being considered for prophylactic brain irradiation (PBI) with no demonstrable intracranial lesions).
* A diagnostic contrast-enhanced magnetic resonance imaging (MRI) demonstrating the presence of 1-6 brain metastases performed within 4 weeks of registration. Note: If small cell lung cancer primary and patient being considered for PBI, MRI must demonstrate no intracranial lesions.
* Patients with totally resected intraparenchymal brain metastases; not all lesions need be resected if all other criteria are satisfied (no more than 6 total lesions)
* The contrast-enhancing intraparenchymal brain tumor must be well circumscribed and must have maximum diameter of no more than 4 cm in any dimension on the enhanced scan. If multiple lesions are present and one lesion is at the maximum diameter, the other(s) must not exceed 3.0 cm in maximum diameter.
* Metastatic lesions must be distributed peripherally, that is, at least 0.5 cm lateral (outside) of the lateral ventricles and/or hippocampus bilaterally. Posterior fossa metastatic lesions are allowed in the study.
* Age 18 years or older.
* Zubrod performance score 0-1.
* Neurologic function score 0, 1, or 2.
* Patients receiving glucocorticoids should be tapered to the lowest possible dose, or altogether, as judged by the participating physician. If glucocorticoid dose is adjusted or given for the first time, patient must remain on stable dose of glucocorticoids for at least 3 days prior to initial Neurocognitive Assessment Protocol (NAP), CT and MR imaging.

Exclusion Criteria:

* Major medical illnesses or psychiatric impairments, which in the investigators opinion will prevent administration or completion of the protocol therapy and/or interfere with follow-up.
* For patients who have undergone subtotal resection, residual disease must be 4 cm in maximum diameter.
* Inability to obtain histologic proof of primary malignancy.
* Patients with leptomeningial metastases documented by MRI or cerebral spinal fluid (CSF) evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S. Anscher, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Massey Cancer Center/Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 08/2007 through 07/2008 in Radiation Oncology clinic
Groups:
- Neural Stem Cell-Preserving Whole Brain RT: Neural Stem Cell-Preserving Whole Brain Radiotherapy
- Standard Whole Brain RT: Standard Whole Brain Radiotherapy
Period: Overall Study
Arm/Group | Neural Stem Cell-Preserving Whole Brain RT | Standard Whole Brain RT
Started | 4 | 4
Completed | 4 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neural Stem Cell-Preserving Whole Brain RT | Standard Whole Brain RT | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (9.7) | 52.0 (0.0) | 59.6 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Secondary Outcome: Increase in the Bi-dimensional Tumor Area for Any of the Tracked Brain Metastases or the Appearance of Any New Brain Metastases on a Follow-up MRI.
Description: Increase in the bi-dimensional tumor area for any of the tracked brain metastases or the appearance of any new brain metastases on a follow-up MRI.
Time Frame: 12 months after end of radiation therapy
Population: Study terminated early due to poor accrual
Groups:
- Standard Whole Brain RT: Standard Whole Brain RT
Arm/Group | Neural Stem Cell-Preserving Whole Brain RT | Standard Whole Brain RT
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Increase in the Bi-dimensional Tumor Area for Any of the Tracked Brain Metastases or the Appearance of Any New Brain Metastases on a Follow-up MRI.
Description: Brain metastases bi-dimensional area
Time Frame: 12 months post RT
Population: Not enough patients were enrolled to allow for any meaningful analysis.
Arm/Group | Neural Stem Cell-Preserving Whole Brain RT | Standard Whole Brain RT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Neural Stem Cell-Preserving Whole Brain RT | Standard Whole Brain RT
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neural Stem Cell-Preserving Whole Brain RT (N=4) | Standard Whole Brain RT (N=4)
Cognitive disturbance - New Brain Mets (Nervous system disorders) | 0 (0) | 1 (1) — Attributed to disease
Neurology - Other (Disease Progression) (Nervous system disorders) | 1 (1) | 0 (0) — Attributed to disease

LIMITATIONS AND CAVEATS:
Trial not completed. Insufficient data to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes